CLINICAL TRIAL: NCT00601822
Title: Cognitive Remediation Therapy for Anorexia Nervosa
Brief Title: Effectiveness of Cognitive Remediation Therapy in Improving Treatment Retention in People With Anorexia Nervosa
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH082706 (NIH); R01MH082706 (NIH); 98328; DATR A2-AID
Record Dates: First submitted 2008-01-04; First posted 2008-01-28 (Estimated); Last update posted 2012-04-10 (Estimated); Status verified 2012-04

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Group receiving cognitive behavioral therapy for anorexia nervosa (CBT-AN)
  Interventions: Behavioral: Cognitive behavioral therapy (CBT)
- 2 (Experimental): Group receiving cognitive behavioral therapy for anorexia nervosa, plus cognitive remediation therapy (CBT-AN+CRT)
  Interventions: Behavioral: Cognitive remediation therapy (CRT); Behavioral: Cognitive behavioral therapy (CBT)

INTERVENTIONS:
Behavioral: Cognitive remediation therapy (CRT) — CRT includes eight sessions over 6 months that aim to improve cognitive flexibility and strengthen thinking skills.
  Arms: 2
Behavioral: Cognitive behavioral therapy (CBT) — CBT includes 20 to 28 weekly psychotherapy sessions over 6 months, depending on treatment group assignment. CBT sessions aim to change participants' beliefs and behaviors toward eating disorders and to teach ways to handle the daily struggles of an eating disorder.

SUMMARY:
This study will evaluate the effectiveness of adding cognitive remediation therapy to cognitive behavioral therapy for treating people with anorexia nervosa.

DETAILED DESCRIPTION:
Anorexia nervosa (AN) is a serious and often chronic eating disorder characterized by low body weight and an obsessive fear of weight gain. People with AN usually try to control body weight by purging, excessive exercise, and/or restrictive eating to near starvation. These dangerous habits and the resultant weight loss in people with AN can lead to serious health complications, including anemia, osteoporosis, and kidney and heart problems. While there is no one known cause for AN, it is believed that a number of psychological, sociological, and neurobiological factors may contribute. Currently, there are no psychological or medication-based treatments known to be highly effective in treating adults with AN. This lack of treatment success may be due to the low retention rates present in AN treatment programs. Cognitive remediation therapy (CRT), a type of psychotherapy that concentrates on improving memory and cognitive flexibility, may be helpful in improving AN treatment adherence. This study will evaluate the effectiveness of adding CRT to cognitive behavioral therapy (CBT) for improving treatment retention rates and for treating people with AN.

Participation in this study will last 1 year and will consist of 6 months of treatment and one follow-up session at 6 months post-treatment. All participants will first undergo baseline assessments, which include interviews and questionnaires about psychological history and AN symptoms, an Eating Disorder Examination (EDE) interview, and a variety of cognitive tests. The questionnaires and cognitive tests will be repeated various times throughout treatment. After baseline assessments, participants will be randomly assigned to receive CBT specifically tailored for AN with or without CRT. Participants assigned to the CBT-only group will receive 28 weekly sessions of CBT with a therapist. Participants assigned to the CBT plus CRT group will receive 8 sessions of CRT and 20 sessions of CBT with a therapist. At each therapy session, participants will have their vital signs checked. In addition, participants will have blood drawn to measure electrolyte levels at baseline and every month during treatment. An electrocardiogram (EKG) will also be taken at baseline and Months 3 and 6. All baseline assessments will be repeated 6 months after the completion of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Meets diagnostic criteria for AN
* Medically stable for outpatient treatment. More information on this can be found in the protocol.
* English literacy

Exclusion Criteria:

* Current psychotic illness
* History of significant brain injury
* Current dependence on drugs or alcohol
* Physical conditions (e.g., diabetes mellitus, pregnancy) known to influence eating or weight
* Previously received CBT or CRT for AN (using the same treatment models as in the study)
* Ideal body weight of less than 75%
* Taking psychotropic medications (antidepressants and antipsychotics) unless on a stable dose for 2 months prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Length of time to discontinue treatment (attrition rate) | Measured at Month 6

SECONDARY OUTCOMES:
Changes in general cognitive processes and those related to anorexia nervosa | Measured at Month 6

CONTACTS AND LOCATIONS:
Overall Officials: James D. Lock, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States